CLINICAL TRIAL: NCT01476488
Title: Conversion of Twice-a-day Tacrolimus to Once-Daily Tacrolimus Extended-Release Formulation in Stable Pediatric Kidney Transplant Recipients
Brief Title: Conversion of Prograf to Advagraf in Pediatric Renal Transplant Recipients
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jongwon Ha, Professor, Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Adva01SNUH
Record Dates: First submitted 2011-07-22; First posted 2011-11-22 (Estimated); Last update posted 2015-05-27 (Estimated); Status verified 2015-05

CONDITIONS: Kidney Transplantation; Pediatric Patients; Maintenance With Tacrolimus
MeSH Terms: interventions — Tacrolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Advagraf (No Intervention): single group, conversion of prograf to advagraf
  Interventions: Drug: tacrolimus

INTERVENTIONS:
Drug: tacrolimus
  Other Names: Prograf; Advagraf

SUMMARY:
This study was designed to compare the pharmacokinetics of Prograf and Advagraf in stable pediatric kidney transplant recipients.

Enrolled patients on prograf will have pharmacokinetic study of tacrolimus for 24 hours and after that, the same dose of advagraf will be prescribed. The patients will have another pharmacokinetic study of tacrolimus after conversion to advagraf.

ELIGIBILITY:
Inclusion Criteria:

* ABO-compatible kidney-only transplantation
* more than 1 year after kidney transplantation
* 5 to 15 years old
* patients maintained on Prograf
* tacrolimus level of determined previously: 4 to 20 ng/ml
* eGFR by Schwartz equation > 50mL/min

Exclusion Criteria:

* patients with acute rejection within 90 days
* patients with acute rejection requiring antibody therapy within 6 months
* patients with more than 2 times of acute rejection within 1 year
* AST/ALT 2 times more than upper normal limit
* ABO-incompatible or crossmatch-positive transplantation
* multiorgan transplantation

Ages: 5 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Dates: Start 2011-07; Primary Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Area Under the Curve of tacrolimus pharmacokinetics (AUC0-24)
  The investigator will compare the changes in AUC0-24 of tacrolimus, Cmax, Tmax and correlation between C0 and Cmax

SECONDARY OUTCOMES:
Number of Participants with Adverse Event

CONTACTS AND LOCATIONS:
Overall Officials: Jongwon Ha, MD, PhD, Principal Investigator — Seoul National University College of Medicine
Locations (1):
- Seoul National University Hospital, Seoul, Seoul, South Korea